CLINICAL TRIAL: NCT06332794
Title: Keep On Keep Up (KOKU4PD) - Developing an App for People With Parkinson's Disease
Brief Title: Keep On Keep Up for Parkinson's
Acronym: KOKU4PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: University of Manchester (Other); Northumbria Healthcare NHS Foundation Trust (Other); Newcastle University (Other); Reason Digital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-2201
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Exercise; Falls prevention; Technology; Physical activity; Co-design
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KOKU user (Experimental): SIngle arm study - all participants will use the KOKU app for 4 weeks.
  Interventions: Device: KOKU4PD

INTERVENTIONS:
Device: KOKU4PD — Exercise at home using the KOKU app for 4 weeks.

SUMMARY:
The goal of this mixed methods, user research study is to evaluate the Keep On Keep Up programme for people with Parkinson's (KOKU4PD).

The main aims of the study are to:

1. To explore the usability and acceptability of the PD specific KOKU programme from a user and health care professional perspective.
2. To produce a KOKU4PD digital program that is ready for National Health Service (NHS) approval and a future effectiveness evaluation.

Participants will use the KOKU4PD app at home for 4 weeks. They will be assessed at baseline and after the 4 weeks to measure aspects of their disease status, mobility, thinking, mood and quality of life. They will also be asked to complete some questionnaires about the usability of the app.

DETAILED DESCRIPTION:
Keep on Keep Up (KOKU) is a digital program available on a tablet that has been designed to engage people in safe and effective falls prevention exercises. KOKU incorporates evidence-based exercise programmes for balance and function and has demonstrated high usability and acceptability in older adults. KOKU is approved by NHS Digital as compliant with regulatory data and safety standards.

Earlier work by the research team has shown that KOKU is effective in improving balance in older adults. However, the effectiveness of KOKU in PD is unknown. The purpose of this study is to explore if app-based exercise is feasible, acceptable and effective in PD, especially in harder-to-reach populations who may not exercise on a regular basis.

Through mixed methods approaches, the proposed study aims to: (i) explore the usability and acceptability of the PD specific KOKU programme from a user and health care professional perspective and (ii) produce a KOKU4PD digital program that is ready for NHS approval and a future effectiveness evaluation.

20 people with PD will be recruited to take part in the study where they will be asked to use the KOKU app independently at home for 4 weeks. A repeated measure design will be employed with assessments performed at the clinical gait lab during two separate sessions lasting between 2-3 hours. Participants will attend the lab for outcomes to be measured at the start and after 4 weeks of exercise with the KOKU app. During the second lab visit, participants will complete a questionnaire about the usability of the KOKU app and take part in an interview to explore their experiences of using it.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's by a movement disorder specialist according to United Kingdom (UK) brain bank criteria (H&Y stage I-III)
* Able to walk and stand without support or assistance from another person
* >40 years
* Stable medication for the previous 1 month and anticipated over a period of 6 months.
* Adequate vision and hearing - to watch and use an iPad or Tablet.Aim: To define the study population/sample

Exclusion Criteria:

* Dementia (<21 on Montreal Cognitive Assessment (MoCA) or as diagnosed according to the Movement Disorder Society guidelines
* Orthopaedic or cardiothoracic ailments that preclude safe walking
* Severe auditory or visual impairment,
* Diagnosis of clinical depression

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Usability of the KOKU app | After 4 weeks of using KOKU at home
  Participants will be asked to complete questionnaires about the usability of the KOKU app and participate in an interview based on their responses to the questionnaires.

SECONDARY OUTCOMES:
Executive clock drawing task (CLOX 1, 2) (mean Change from baseline) | After 4 weeks of using KOKU at home
  A clock drawing task (CLOX) designed to elicit executive impairment and discriminate it from non-executive constructional failure.
Trail Making Test (mean Change from baseline) | After 4 weeks of using KOKU at home
  Timed written test of visual function and scanning
Freezing of Gait Questionnaire (mean Change from baseline) | After 4 weeks of using KOKU at home
  Self-report questionnaire
Falls Efficacy scale (mean Change from baseline) | After 4 weeks of using KOKU at home
  Self-report questionnaire (minimum 16 (no concern about falling) to maximum 64 (severe concern about falling)
Parkinson's disease quality of life questionnaire - PDQ-39 (mean Change from baseline) | After 4 weeks of using KOKU at home
  The 39 item questionnaire offers a patient reported measure of health status and quality of life. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100 (100 = more health problems).
Mini-BESTest (mean Change from baseline) | After 4 weeks of using KOKU at home
  The Mini-BESTest is a clinical balance test that has shown a high sensitivity in detecting balance impairments in elderly people with Parkinson's disease. The Mini- BESTest consists of 14 items, with a maximum (best) score of 28 points.
Two minute walk test, single and dual task (mean Change from baseline) | After 4 weeks of using KOKU at home
  Participant walks continually for 2 minutes; for dual task, participant is asked to recall numbers as they are walking
EuroQol-5 Dimension Quality of Life tool - EQ5D-5L (mean Change from baseline) | After 4 weeks of using KOKU at home
  Self-report quality fo life questionnaire - EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state.
Activities-specific Balance Confidence (ABC) Scale (mean Change from baseline) | After 4 weeks of using KOKU at home
  The Activities-specific Balance confidence (ABS) scale is a questionnaire developed to assess older individual's balance confidence in performing daily activities. There are 16 items, representing daily activities. Participants are asked to answer, with a score from 0% (not confident at all) to 100% (completely confident) in increments of 10%, how confident they are in performing each activity. The average score obtained is an indication on balance confidence.
  A score of > 80% indicates high level of functioning. A score of 50%-80% indicates moderate level of functioning. A score of < 50% indicates low levels of functioning. Additionally, a score of < 67% suggests substantial risk of falling.
Multidimensional Fatigue Inventory (MFI) (mean Change from baseline) | After 4 weeks of using KOKU at home
  The MFI is a 20-item inventory scored on a 5-point Likert scale and measures five dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. The MFI dimension scores range from 4 to 20 (most severe) and have been credited with reliably measuring fatigue severity in each dimension.
Technology Acceptance questionnaire | After 4 weeks of using KOKU at home
  Self-report questionnaire, based on the Technology Acceptance Model. There are 15 items which participants have to rate on a scale of 1 (= strongly disagree) to 7 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will only be available to members of the study team.